CLINICAL TRIAL: NCT03224260
Title: Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety and Pharmacokinetics of BMS-986177 in Healthy Japanese Participants
Brief Title: To Evaluate the Safety and Pharmacokinetics of BMS-986177 in Healthy Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: CV010-011
Record Dates: First submitted 2017-07-18; First posted 2017-07-21 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — milvexian

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): Receive 50 mg BMS-986177 once daily or placebo
  Interventions: Drug: BMS-986177; Other: Matched Placebo
- Treatment B (Experimental): Receive 200 mg BMS-986177 once daily or placebo
  Interventions: Drug: BMS-986177; Other: Matched Placebo
- Treatment C (Experimental): Receive 500 mg BMS-986177 once daily or placebo
  Interventions: Drug: BMS-986177; Other: Matched Placebo

INTERVENTIONS:
Drug: BMS-986177 — Oral Suspension
Other: Matched Placebo — Oral Suspension

SUMMARY:
Access the safety, tolerability, and pharmacokinetics of BMS-986177 in healthy Japanese participants after multiple doses are administered.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be first-generation Japanese (born in Japan and not living outside of Japan for > 10 years; both parents must be ethnically Japanese)
* Body Mass Index 18.0 to 25.0 kg/m2, inclusive
* Women must not be of nonchildbearing potential (cannot become pregnant)

Exclusion Criteria:

* Any significant acute or chronic medical illness
* History of allergy to BMS-986177 or other factor Xia inhibitors and/or formulation excipients or history of any significant drug allergy (such as anaphylaxis or hepatotoxicity)
* History or evidence of abnormal bleeding or coagulation disorder

Other protocol defined inclusion and exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of Death | 30 days after last dose
  Measured by investigator assessment
Incidence of Serious Adverse Events (SAEs) | 30 days after last dose
  Measured by investigator assessment
Incidence of Adverse Events (AEs) Leading to Discontinuation of Study Therapy | 17 days
  Measured by investigator assessment
Incidence of Adverse Events (AEs) Resulting in Clinically Significant Bleeding | 17 days
  Measured by investigator assessment
Changes in Vital Signs (heart rate, systolic blood pressure, diastolic blood pressure, respiration rate, and temperature) | 17 days
  Measured by investigator assessment
Change from baseline in electrocardiogram findings (ECGs) | 17 days
  Measured by investigator assessment

CONTACTS AND LOCATIONS:
Locations (1):
- West Coast Clinical Trials, Anaheim, California, United States

REFERENCES:
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/recalls/
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS clinical trial educational resource — https://www.bmsstudyconnect.com/s/US/English/USenHome